CLINICAL TRIAL: NCT05927649
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, 3-Way Crossover Study in Healthy Subjects to Determine the Effect of Omaveloxolone on QTc Interval
Brief Title: A TQTc Study for Omaveloxolone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Celerion (Industry); Q2 Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 408-C-2201
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Health Adult Subjects
Keywords: C-QTc; omaveloxolone; TWTc; moxifloxacin
MeSH Terms: interventions — omaveloxolone; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence ABC (Experimental): Subjects receive three treatments (A: omaveloxolone 450 mg, B: omaveloxolone matching placebo 450 mg and C: moxifloxacin 400 mg) administered in a single dose with the standard FDA high-fat meal in three periods. Treatment A (Period 1 from Day 1 - 15), Treatment B (Period 2 from Day 15 - 29), and Treatment C(Period 3 from Day 29 -32)
  Interventions: Drug: Omaveloxolone; Drug: Moxifloxacin
- Sequence BAC (Experimental): Subjects receive three treatments (A: omaveloxolone 450 mg, B: omaveloxolone matching placebo 450 mg and C: moxifloxacin 400 mg) administered in a single dose with the standard FDA high-fat meal in three periods. Treatment B (Period 1 from Day 1-15), Treatment A (Period 2 from Day 15 - 29, and Treatment C (Period 3 from Day 29 to 32)
  Interventions: Drug: Omaveloxolone; Drug: Moxifloxacin
- Sequence ACB (Experimental): Subjects receive three treatments (A: omaveloxolone 450 mg, B: omaveloxolone matching placebo 450 mg and C: moxifloxacin 400 mg) administered in a single dose with the standard FDA high-fat meal in three periods. Treatment A (Period 1 from Day 1-15), Treatment C (Period 2 from Day 15 -18), and Treatment B (Period 3from Day 18 - 32)
  Interventions: Drug: Omaveloxolone; Drug: Moxifloxacin
- Sequence BCA (Experimental): Subjects receive three treatments (A: omaveloxolone 450 mg, B: omaveloxolone matching placebo and C: moxifloxacin 400 mg) administered in a single dose with the standard FDA high-fat meal in three periods. Treatment B (Period 1 from Day 1 - 15), Treatment C (Period 2 from Day 15 to 18), and Treatment A (Period 3 from Day 18 - 32)
  Interventions: Drug: Omaveloxolone; Drug: Moxifloxacin
- Sequence CAB (Experimental): Subjects receive three treatments (A: omaveloxolone 450 mg, B: omaveloxolone matching placebo and C: moxifloxacin 400 mg) administered in a single dose with the standard FDA high-fat meal in three periods. Treatment C (Period 1 from Day 1 - 4), Treatment A (Period 2 from Day 4 - 18), and Treatment B (Period 3 from Day 18 - 32)
  Interventions: Drug: Omaveloxolone; Drug: Moxifloxacin
- Sequence CBA (Experimental): Subjects receive three treatments (A: omaveloxolone 450 mg, B: omaveloxolone matching placebo and C: moxifloxacin 400 mg) administered in a single dose with the standard FDA high-fat meal in three periods. Treatment C (Period 1 from Day 1 - 4), Treatment B (Period 2 from Day 4 - 18), and Treatment A (Period 3 from Day 18 - 32)
  Interventions: Drug: Omaveloxolone; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Omaveloxolone — Omaveloxolone capsules
  Other Names: RTA 408
Drug: Moxifloxacin — Moxifloxacin capsules

SUMMARY:
This is a randomized, double blind, placebo and active (moxifloxacin open label) controlled study in healthy subjects to assess the effect of the supratherapeutic exposure of omaveloxolone on QTc interval. Moxifloxacin will be used as an active control and will be administered as open label. Omaveloxolone and placebo will be administered in a blinded fashion. All treatments will be administered after an FDA high-fat meal. Concentration-QTc (C-QTc) analysis is the primary analysis for the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and/or females, 18 to 55 years of age (inclusive) at the time of screening.
* BMI at screening between 18.0 and 32.0 kg/m2 (inclusive)
* Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

* History of clinically significant drug allergies, including allergies to any of the components of the study drugs (omaveloxolone and moxifloxacin) and/or clinically significant food allergies as determined by the investigator.
* Subject has an ECG abnormality, including corrected QT interval (QTc)> 450 msec for males, and > 460 msec for females, HR < 45 bpm or > 100 bpm after 5 minutes in supine position, PR interval > 220 msec, or QRS interval > 110 msec.
* Subject has allergy to band aids, adhesive dressing, or medical tape.
* Subject has hypotension (systolic blood pressure blood pressure [BP] ≤ 90 mmHg, diastolic BP ≤ 50 mmHg), or hypertension (systolic BP ≥ 140 mmHg, diastolic BP ≥ 90 mmHg) at screening.
* Subject has history of prolonged QTc, cardiac arrhythmia, or first-degree relatives with congenital Long QT syndrome or unexplained sudden death in young age.
* Subject has a history of unstable angina, syncope, coronary artery disease, myocardial infarction, congestive heart failure (CHF), transient ischemic attack (TIA), or neurological disorder.
* Presence or history of any significant cardiovascular, gastrointestinal, hepatic, renal, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease, as determined by the investigator.
* Presence of any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines.
* Requirement for any over the counter and/or prescription medication, vitamins, and/or herbal supplements on a regular basis
* Use of any medications (over the counter and/or prescription medication), vitamins, and/or herbal supplements, within the 14-days prior to study drug administration or within 5 halflives (if known), whichever is longer
* History of drug or alcohol abuse in the last 6 months as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition.
* Positive test result for drugs of abuse, alcohol, or cotinine at screening or Day -1.
* Positive test result for hepatitis B surface antigen, hepatitis C virus antibodies, or HIV antibodies at screening.
* Positive test result for COVID-19 at Day -1.
* Blood donation (excluding plasma donation) of approximately 500 mL within 56 days before screening or plasma donation within 7 days before screening.
* Receipt of any investigational product within a time period equal to 10 half-lives of the product, if known, or a minimum of 30 days before study drug administration.
* Consumption of alcohol within 72 hours before study drug administration.
* Consumption of grapefruit, grapefruit products, star fruit, star fruit products, Seville oranges, or Seville orange products within the 72-hour period before study drug administration.
* Use of tobacco or nicotine-containing products within the 6-month period preceding study drug administration.
* Current enrollment in another clinical study.
* Previous enrollment in any clinical study involving omaveloxolone.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in placebo-corrected QTcF (∆∆QTcF) | At Day 1 of each period, which is 14 days for both Treatment A and Treatment B and 4 days for Treatment C
  The relationship between ∆QTcF and omaveloxolone and its metabolites, M17 and M22 plasma concentrations will be investigated by a linear mixed effects modeling approach with ∆ QTcF as the dependent variable, time-matched concentration of omaveloxolone and its metabolites as a continuous covariate (ie, 0 for placebo), and centered baseline QTcF as an additional covariate, treatment (active = 1; or placebo = 0) and time as categorical factors, and a random intercept and slope per subject.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Valentine, DO, Principal Investigator — Celerion
Locations (1):
- Celerion, Inc., Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/